CLINICAL TRIAL: NCT01921413
Title: Clinical Validation of Fyodor Urine Malaria Test (UMT)
Brief Title: Clinical Performance Evaluation of Fyodor Urine Malaria Test (UMT)
Status: Completed | Type: Observational
Sponsor: Fyodor Biotechnologies Inc (Industry)
Collaborators: University of Lagos, Nigeria (Other); Johns Hopkins University (Other); Federal Ministry of Health, Nigeria (Other Government); Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: UMT Evaluation
Record Dates: First submitted 2013-08-07; First posted 2013-08-13 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; Clinical Malaria; Fever; Schistosoma hematobium; Rheumatoid arthritis
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Fever; Schistosomiasis haematobia; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Urine Malaria Test — Rapid non-invasive malaria diagnostic test
  Other Names: UMT

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the one-step Fyodor Urine Malaria Test (UMT), to determine its accuracy (sensitivity and specificity) for the diagnosis of Plasmodium falciparum malaria in febrile patients. A total of 1500 properly consented children and adults presenting with fever (axillary temperature ≥37.5°C) or history of fever in the last 48 hours (Group 1), 250 apparently "healthy" individuals (Control, Group 2), and 50 patients with Schistosoma hematobium and Rheumatoid arthritis (Group 3), will be recruited. Matched urine and fingerprick (capillary) blood samples will be collected and tested using the UMT and, Binax NOW® malaria rapid diagnostic test (blood test) and thick smear microscopy, respectively. The overall agreement of the UMT results to the Binax NOW analysis and thick smear microscopy will be used to establish UMT sensitivity and specificity.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the clinical performance (sensitivity and specificity) of Fyodor UMT for detecting Plasmodium falciparum malaria in febrile patients.

Secondary Objectives:

* To monitor time-to-clearance of the cognate parasite protein from patient urine
* To assess the potential effects of proteinuria, inflammation and anti-fever medications on Fyodor UMT performance
* To determine UMT performance when used for asymptomatic (afebrile) individuals, who may be carriers of the parasite.

Study Design:

* Randomized, multi-center clinical study
* Participants will be recruited from primary healthcare centers across four local government areas in Lagos State, and two schistosomiasis communities in Abeokuta-North Local Government Area of Ogun State, both in southwest Nigeria
* 1500 participants (comprising children aged 2-14 years and adults of both genders) with fever (axillary temperature ≥37.5°C) or recent history of fever in the last 48 hours (Group 1), 250 apparently "healthy" individuals (Control, Group 2), and 50 patients with Schistosoma hematobium and Rheumatoid arthritis (Group 3), will be recruited
* Binax NOW RDT-positive patients will be treated for malaria infection with Artesunate-Amodiaquine or Dihydroartemisinin-Piperaquine Sulphate, following national treatment policy
* To assess if the UMT target antigen persists in urine after treatment, 100 treated Group 1 participants with both Binax NOW and UMT positive results will be randomly selected and followed up on days 3, 7, 14, 21, and 28, using an adaptation of the WHO (2009) Protocol for Drug Therapeutic Efficacy Assessments (http://whqlibdoc.who.int/publications/2009/9789241597531_eng.pdf)
* To test the clinical specificity of the UMT, active recruitment will include 250 individuals of both genders with asymptomatic P. falciparum malaria infection (apparently "healthy, normal control group 2), and 50 with Schistosoma haematobium infection and/or rheumatoid arthritis (Group 3) - two unrelated medical conditions known to elicit proteinuria in patients (Lehman et al., 1975; Adebajo et al., 1994; Tighe & Carson, 1997)
* Participants with elevated Rheumatoid Factor (RF+) test result (i.e. RF >60 u/mL or >1:80 liter) are associated with severe rheumatoid disease. Schistosoma haematobium infection is confirmed by microscopy with egg identification or by serology
* This 6-month study will be implemented July-December 2013, during both rainy and dry seasons when malaria transmission is high and low, respectively.

Study Area:

The study will be coordinated by The ANDI Center of Excellence for Malaria Diagnosis - an International Malaria Microscopy Training & RDT Quality Assurance Testing center, & a WHO/TDR/FIND Malaria Specimen Bank Site at the College of Medicine, The University of Lagos. It will be conducted in seven primary healthcare facilities across four local government areas in Lagos State. Lagos State is situated in the southwestern part of Nigeria, and made up of densely populated urban areas and sprawling suburban areas. Malaria transmission occurs throughout the year with periods of intense seasonal malaria transmission during the rainy season. Temperatures are usually high and water pools created during the rainy season provide breeding sites for the malaria vectors, leading to epidemic outbreaks with high morbidity rates. The state is endemic for malaria, with peak transmission between April-September.

The sampling for Schistosomiasis will be carried out in Imalodo and Abuletutu schistosomiasis communities in Abeokuta-North Local Government Area of Ogun State, also in southwest Nigeria.

Description of the Study Design:

The specific aims of the study are to determine the clinical sensitivity and specificity of the UMT, and to establish assay performance characteristics in healthy asymptomatic volunteers, compared to blood smear microscopy, and Binax NOW test (Predicate device). A total of 1,800 participants, comprising children and adults of both genders presenting with malaria-like fever symptoms, patients with unrelated medical conditions (Schistosoma hematobium infection and rheumatoid arthritis, as well as apparently "healthy" (asymptomatic) control individuals will be enrolled. Febrile patients with malaria-like symptoms will be enrolled during both the rainy and dry seasons, yielding field samples during periods of both high and low malaria transmission.

Matched urine and fingerprick blood samples will be collected and tested using the UMT, and Binax NOW and microscopy, respectively. Urine and blood testing with the UMT and Binax NOW, respectively, will be performed on-site in a blinded fashion. Each urine sample will also be tested using a urinalysis dipstick and its' physicochemical characteristics (pH, protein, sugar, specific gravity, etc) are recorded. Two thin and thick blood smear slides (prepared on the same slide) per participant will be prepared from the blood specimen. One slide will be independently read by two microscopists at the ANDI Center of Excellence for Malaria Diagnosis, an internationally reputed training and referral center for malaria microscopy. The second slide will be archived for future quality assurance purpose, and thereafter shipped to Fyodor along with the remaining urine samples. Per convention, microscopic reading of blood smears will be used as the gold standard for malaria diagnosis. Patients testing positive with Binax NOW will be treated with Artesunate-Amodiaquine or Dihydroartemisinin-Piperaquine Sulphate. No clinical decision will be made based on the UMT results alone. Nevertheless, the standard routine malaria diagnostic tests will be used to manage the patient in the facility where they present. The overall agreement of the UMT and Binax NOW to microscopy analysis will be used to establish UMT sensitivity, specificity, and substantial equivalence/non-inferiority to Binax NOW test.

UMT Test Procedure:

* Add 200 µl of the freshly collected urine into a 1.5 ml or 2 ml test tube immediately before testing
* Dip the UMT strip into the urine sample and allow sample to wick up and saturate the strip for 10 minutes
* Remove the strip from the urine specimen, and place on its foil pouch packaging
* Allow reaction to proceed for 20 minutes
* Record result as positive (POS; both Test and Control Lines appear), negative (NEG; only the Control Line appears) or invalid (INV; Control Line does not appear).

Study Quality Assurance:

This study will be conducted in accordance with good clinical practices.

* Site training: All investigators, technicians and research staff working on this UMT study will be trained and certified in the conduct of studies involving human subjects per ICH guidelines
* Site Visits: Site monitoring visits will be conducted according to the guidelines outlined in the study protocol
* Blinding of Results: Separate teams will be organized to conduct patient enrollment, laboratory (Binax NOW) testing, diagnostic microscopy, data entry, and data analysis
* Control UMT Testing: Known positive and negative control materials will be used to verify UMT performance on a daily basis
* Data Collection: Research staff will fill out all data collection forms at each visit, even if a participant has not had all of the tests completed; missed follow up visits will be documented, as appropriate, on the case report forms
* The Study Coordinator will manage field research staff and provide administrative support at study sites on a day-to-day basis
* Study Quality Assurance Coordinator is qualified by training and experience, and will monitor the conduct of the trial to ensure compliance with the approved study protocol.

This clinical study will be conducted in accordance with the study protocol as approved by the Research Grants & Experimentation Ethics Committee of the College of Medicine University of Lagos, Nigeria, the Nigerian Health Research Ethics Committee guidelines, the ICH Harmonised Tripartite Guideline for Good Clinical Practice and 45CFR46 and 21CFR50, the WHO-FIND-CDC Malaria RDT Product Testing Methods Manual (Version 3), the abbreviated or non-significant risk provision of the Investigational Device Exemptions (IDE) Regulations (21 CFR Part 812.2(b)), the Protection of Human Subjects Regulations, including Subpart B Informed Consent of Human Subjects (21 CFR Part 50), the Institutional Review Board Regulations (21 CFR Part 56); and, the Financial Disclosure by Clinical Investigators Regulations (21 CFR Part 54).

ELIGIBILITY:
Inclusion Criteria:

Group 1 - Febrile Patients:

* Age: two years or older
* Fever at the time of presentation (axillary temperature ≥37.5°C), or history of fever within the past 48 hours
* Subjects with concurrent illnesses not listed in the exclusion criteria will be evaluated and treated for these illnesses and included in the study
* Written informed consent obtained from the participant or parent/guardian

Group 2 - Apparently Healthy Individuals:

* Children 2 years or older, as well as adults of both genders
* Afebrile
* No history of fever within the past 48 hours
* Negative Binax NOW test confirmed by Negative blood smear for clinical malaria

Group 3 - Patients with unrelated medical conditions known to elicit proteinuria in patients:

* Children 2 years or older, as well as adults
* Afebrile
* No history of fever within the past 48 hours
* Negative Binax NOW test confirmed by Negative blood smear for clinical malaria

Exclusion Criteria:

* Pregnancy
* Patients with respiratory distress, diffuse bleeding, recent seizures, coma, inability to drink, persistent vomiting, or prostration
* Chronic use of a medication (such as trimethoprim-sulfamethoxazole for preventing AIDS-associated opportunistic infections) with known antimalarial activity
* Any condition that in the opinion of the Principal Investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will comprise of individuals 2 years or older of both genders with fever (axillary temperature ≥37.5°C) (Group 1), apparently "healthy" individuals (Control, Group 2), and patients positive for Rheumatoid factor (Group 3), will be recruited will be recruited at primary healthcare facilities across four local government areas in Lagos State, southwest Nigeria - Ikorodu, Surulere, Shomolu and Ibeju-Lekki. The sampling for Schistosomiasis will be carried out in Imalodo and Abuletutu communities in Abeokuta-North Local Government Area of Ogun State, also in southwest Nigeria.
Sampling Method: Probability Sample
Enrollment: 1893 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of the UMT for Clinical Malaria Diagnosis | Acute (day 0) fever suspected of being malaria or recent history of fever in the past 48 hours
  • Establish sensitivity and specificity of the UMT for malaria diagnosis in febrile patients.

SECONDARY OUTCOMES:
Monitoring the Effectiveness of Malaria Treatment by Rapid Urine Testing | From Day 3 of ACT administration, and followed up weekly for 28 days
  * Determine how quickly the cognate malaria antigens are cleared from patient urine after the prescribed three-day course of artemisinin-combination therapy (ACT);
  * Negative UMT results (as confirmed by microscopy during the study) will establish the effectiveness of malaria treatment and provide a means to rapidly monitor effective treatment;
  * Establish broader UMT utility for epidemiological monitoring in asymptomatic (afebrile) individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Wellington A Oyibo, PhD, Principal Investigator — ANDI Centre of Excellence for Malaria Diagnosis, International Malaria Microscopy Training & RDT QA Center, & WHO/TDR/FIND Malaria Specimen Bank Site, Department of Medical Microbiology & Parasitology, College of Medicine, University of Lagos, Nigeria; William (Bill) Brieger, DrPH, Study Director — Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland, USA; Wendy O'Meara, PhD, Study Director — Duke University School of Medicine, Durham, North Carolina, USA; Nnenna Ezeigwe, MBBS, FMCPH, Study Director — Coordinator, National Malaria Control Program/Federal Ministry of Health, Abuja, Nigeria; Godwin Ntadom, MBBS, MPH, Study Director — Head, Case Management, National Malaria Control Program/Federal Ministry of Health, Abuja, Nigeria
Locations (1):
- College of Medicine of the University of Lagos, Idi Araba, Lagos, Nigeria

REFERENCES:
- [Background] Adebajo AO, Cawston TE, Hazleman BL. Rheumatoid factors in association with rheumatoid arthritis and infectious diseases in West Africans. J Rheumatol. 1994 May;21(5):968-9. No abstract available. PMID 8064747
- [Background] Tighe H, Warnatz K, Brinson D, Corr M, Weigle WO, Baird SM, Carson DA. Peripheral deletion of rheumatoid factor B cells after abortive activation by IgG. Proc Natl Acad Sci U S A. 1997 Jan 21;94(2):646-51. doi: 10.1073/pnas.94.2.646. PMID 9012838
- [Background] Lehman JS Jr, Mott KE, De Souza CA, Leboreiro O, Muniz TM. The association of Schistosomiasis mansoni and proteinuria in an endemic area. A preliminary report. Am J Trop Med Hyg. 1975 Jul;24(4):616-8. doi: 10.4269/ajtmh.1975.24.616. PMID 1155697